CLINICAL TRIAL: NCT07340970
Title: Patient Perception of Sensory Stimuli During Elective Cesarean Delivery Under Neuraxial Anesthesia (PIONEER)
Brief Title: Sensory Stimuli During Cesarean Delivery
Acronym: PIONEER
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Juliana Barrera, Clinical Asisstant Professor, University of British Columbia
Other Study IDs: H25-02656
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Intraoperative Pain
Keywords: cesarean delivery; neuraxial anesthesia; intraoperative pain; intraoperative sensation; peritraumatic distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort: Healthy patient undergoing elective cesarean delivery under neuraxial anesthesia
  Interventions: Other: Standardized intraoperative and postoperative patient-reported assessments

INTERVENTIONS:
Other: Standardized intraoperative and postoperative patient-reported assessments — Brief patient self-assessments at six intraoperative time points (questions + VAS + diagram), and postoperative questionnaires (PDI, EPDS, PCL-5) through 6 months postpartum.

SUMMARY:
This study will follow people having a planned cesarean birth with a spinal or combined spinal-epidural anesthetic. The investigators will ask what kinds of sensations participants feel during the operation, how often these happen, and whether any of the sensations feel as unacceptable or too uncomfortable.

Participants will be asked a few short questions at six set times during the surgery. Participants will also complete short questionnaires before surgery and again after birth (up to 6 months) to help us understand mood, stress, and overall wellbeing.

DETAILED DESCRIPTION:
Cesarean delivery is common and neuraxial anesthesia is the standard technique; however, a meaningful proportion of patients experience intraoperative pain or distressing sensations. Existing research often relies on retrospective recall, surrogate markers (e.g., medication use), and variable definitions of intraoperative pain, with limited prospective characterization of the sensory experiences that patients perceive and whether participants interpret them as painful or otherwise unacceptable.

PIONEER is a prospective, longitudinal cohort study enrolling healthy pregnant patients undergoing elective cesarean delivery at BC Women's Hospital. The primary objective is to estimate the incidence of intraoperative sensory stimuli that are self-reported as unacceptable (i.e., sensations the participant reports as unacceptable and needing treatment). Intraoperative data will be collected at six defined surgical milestones from block confirmation to skin closure via short patient questions. Postoperative and longitudinal follow-up will assess postpartum distress, depression, and PTSD symptoms. Clinical care is not directed by the study; anesthetic and surgical management remains at the discretion of the treating team.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant patients ≥36 weeks gestational age
* ASA Physical Status Class 2-3
* Elective cesarean delivery
* Age ≥19 years
* English-speaking

Exclusion Criteria:

* Known history of chronic pain or pain disorders
* Currently taking medications with analgesic properties
* Known history of neurological conditions that may impair normal sensation
* Cesarean delivery requiring epidural top-up or de novo general anesthesia

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy pregnant patients ≥36 weeks gestational age undergoing elective cesarean delivery under neuraxial anesthesia at BC Women's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative sensory stimuli perceived as unacceptable | From date of enrollment until the date of cesarean delivery completed, assessed up to 1day.
  Proportion of participants who report experiencing any intraoperative sensory stimulus that they subjectively self-report as unacceptable.

SECONDARY OUTCOMES:
Qualitative description of unacceptable sensory stimuli | From date of enrollment until the date of cesarean delivery completed, assessed up to 1day.
  Thematic categorization of participant responses
Severity of intraoperative sensory stimuli | From date of enrollment until the date of cesarean delivery completed, assessed up to 1day.
  Sensation intensity rated using a 0-10 visual analog scale (VAS) at each intraoperative assessment time point.
Total intraoperative supplemental IV analgesia received | From date of enrollment until the date of cesarean delivery completed, assessed up to 1day.
  Total dose(s) of supplemental IV analgesic medications administered intraoperatively, abstracted from the medical record/anesthesia record.
PTSD symptoms over time | From date of enrollment until the date of follow-up completion, assessed up to 6 months post-partum.
  PTSD Checklist for DSM-5 (PCL-5) score measured longitudinally.
Depressive symptoms over time | From date of enrollment until the date of follow-up completion, assessed up to 6 months post-partum.
  Edinburgh Postnatal Depression Scale (EPDS) score measured longitudinally.
Peritraumatic distress over time | From date of enrollment until the date of follow-up completion, assessed up to 6 months post-partum.
  Peritraumatic Distress Inventory (PDI) score measured longitudinally.
Postoperative pain intensity (NRS) | From date of enrollment until the date of discharge from hospital, assessed up to 3 weeks post-partum.
  0-10 Numerical Rating Scale (NRS) pain scores collected during the first 48 hours of admission, per clinical charting.
In-hospital opioid requirement (MME) | From date of enrollment until the date of discharge from hospital, assessed up to 3 weeks post-partum.
  Total opioid dose administered from end of surgery until hospital discharge, converted to oral morphine milligram equivalents (MME).

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Kruthof, MD, MSc, FRCPC, Principal Investigator — Department of Anesthesia BC Women's Hospital
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saulnier L, Chau A, Barrera J, Massey S. Influence of Planned Versus Unplanned Cesarean Delivery on Postpartum Peritraumatic Distress: A Prospective Observational Study. J Obstet Gynaecol Can. 2025 Nov;47(11):103114. doi: 10.1016/j.jogc.2025.103114. Epub 2025 Sep 10. PMID 40939978
- [Background] Jagodnik KM, Ein-Dor T, Chan SJ, Titelman Ashkenazy A, Bartal A, Barry RL, Dekel S. Screening for post-traumatic stress disorder following childbirth using the Peritraumatic Distress Inventory. J Affect Disord. 2024 Mar 1;348:17-25. doi: 10.1016/j.jad.2023.12.010. Epub 2023 Dec 7. PMID 38070747
- [Background] Stanford SER. What is 'genuine' failure of neuraxial anaesthesia? Anaesthesia. 2022 May;77(5):523-526. doi: 10.1111/anae.15723. Epub 2022 Mar 25. No abstract available. PMID 35332526
- [Background] Mehdiratta JE, Saab R, Chen Z, Li YJ, Habib AS. Patient and procedural risk factors for increased postoperative pain after cesarean delivery under neuraxial anesthesia: a retrospective study. Int J Obstet Anesth. 2020 Nov;44:60-67. doi: 10.1016/j.ijoa.2020.07.006. Epub 2020 Jul 21. PMID 32799069
- [Background] Plaat F, Stanford SER, Lucas DN, Andrade J, Careless J, Russell R, Bishop D, Lo Q, Bogod D. Prevention and management of intra-operative pain during caesarean section under neuraxial anaesthesia: a technical and interpersonal approach. Anaesthesia. 2022 May;77(5):588-597. doi: 10.1111/anae.15717. Epub 2022 Mar 24. PMID 35325933
- [Background] Stanford SE, Bogod DG. Failure of communication: a patient's story. Int J Obstet Anesth. 2016 Dec;28:70-75. doi: 10.1016/j.ijoa.2016.08.001. Epub 2016 Aug 23. PMID 27717633
- [Background] Lopez U, Meyer M, Loures V, Iselin-Chaves I, Epiney M, Kern C, Haller G. Post-traumatic stress disorder in parturients delivering by caesarean section and the implication of anaesthesia: a prospective cohort study. Health Qual Life Outcomes. 2017 Jun 2;15(1):118. doi: 10.1186/s12955-017-0692-y. PMID 28577570
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Landau R, Richebe P. Tailoring postoperative pain management with a procedure-specific approach: how to best apply this concept to caesarean deliveries. Anaesthesia. 2021 May;76(5):587-589. doi: 10.1111/anae.15251. Epub 2020 Oct 14. No abstract available. PMID 33280087
- [Background] Charles EA, Carter H, Stanford S, Blake L, Eley V, Carvalho B, Sultan P, Kua J, O'Carroll JE. Intraoperative Pain during Cesarean Delivery under Neuraxial Anesthesia: A Systematic Review and Meta-analysis. Anesthesiology. 2025 Jul 1;143(1):156-167. doi: 10.1097/ALN.0000000000005486. Epub 2025 Apr 4. PMID 40184602
- [Background] Frank E, Sharpe EE, Kohn G, Kohl-Thomas B, Shaver C, Hofkamp MP. Predictors of intraoperative pain during cesarean delivery under regional anesthesia. Proc (Bayl Univ Med Cent). 2022 Jun 14;35(5):595-598. doi: 10.1080/08998280.2022.2086789. eCollection 2022. PMID 35991734
- [Background] Sanchez J, Prabhu R, Guglielminotti J, Landau R. Pain during cesarean delivery: A patient-related prospective observational study assessing the incidence and risk factors for intraoperative pain and intravenous medication administration. Anaesth Crit Care Pain Med. 2024 Feb;43(1):101310. doi: 10.1016/j.accpm.2023.101310. Epub 2023 Oct 20. PMID 37865217